CLINICAL TRIAL: NCT01023971
Title: Study of Macular Function During Anti-VEGF Treatment
Brief Title: Macular Function During Anti-VEGF Treatment
Acronym: MAFAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Liverpool University Hospital (Other Government)
Responsible Party: Simon P Harding, Royal Liverpool University Hospital
Other Study IDs: Trust R&D_3704
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Patients investigated with mfERG and MP-1
- Group B: Patients investigated by Laser Doppler Flowmetry

SUMMARY:
The purpose of this study is to determine the changes in macular function during anti-VEGF treatment for neovascular age-related macular degeneration.

DETAILED DESCRIPTION:
Macular function will be investigated using visual acuity, contrast sensitivity, mfERG and microperimetry.

ELIGIBILITY:
Inclusion Criteria:

* Neovascular AMD in first or second eyes
* angiographic signs of active subfoveal or juxtafoveal choroidal neovascularization (CNV)
* BCVA ≥35 ETDRS letters

Exclusion Criteria:

* Spherical equivalent ≥ ± 6 D
* Previous treatments for CNV in the studied eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMD clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-01

PRIMARY OUTCOMES:
mfERG central ring amplitude density | 12 months

SECONDARY OUTCOMES:
Mean retinal sensitivity (dB) in three concentric rings (4°, 8° & 12°) | 12 months
Choroidal blood flow (ChBFlow) at fovea and at optic nerve head | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon P HARDING, FRCOphth, MD, Principal Investigator — University of Liverpool
Locations (1):
- Clinical Eye Research Centre, Liverpool, United Kingdom

REFERENCES:
- [Derived] Campa C, Hagan R, Sahni JN, Brown MC, Beare NA, Heimann H, Harding SP. Early multifocal electroretinogram findings during intravitreal ranibizumab treatment for neovascular age-related macular degeneration. Invest Ophthalmol Vis Sci. 2011 Jun 1;52(6):3446-51. doi: 10.1167/iovs.10-6588. PMID 21357390